CLINICAL TRIAL: NCT06442020
Title: Low Intensity Shock Wave Therapy in the Rehabilitation Treatment of Erectile Dysfunction After Robotic Radical Prostatectomy: Randomized Controlled Trial
Brief Title: Low Intensity Shock Wave Therapy in the Rehabilitation Treatment of Erectile Dysfunction After Robotic Radical Prostatectomy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RS1874/23
Record Dates: First submitted 2024-03-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP 1: LiESWT in association with PDE5i (Experimental): Therapeutic association between low intensity extracorporeal shock waves LiESWT and the early introduction of the phosphodiesterase 5 inhibitor PDE5i
  Interventions: Procedure: Tadalafil (PDE5i)
- GROUP 2: PDE5i alone (Active Comparator): Control group, administration of the phosphodiesterase 5 inhibitor PDE5i, as per clinical practice
  Interventions: Procedure: Tadalafil (PDE5i)

INTERVENTIONS:
Procedure: Tadalafil (PDE5i) — Tadalafil at a dose of 5mg/day

SUMMARY:
The study deals with the hypothesis that LiESWT in addition to the administration of PDE5i can improve sexuality rehabilitation with faster recovery of a valid erection and higher IIEF-5 scores in the short and medium-term follow-up.

DETAILED DESCRIPTION:
Prospective randomized controlled trial (RCT) designed to provide high level evidences describing the role of Low-intensity Extracorporeal Shock Wave Therapy LiESWT plus early introduction of PDE5i vs early PDE5i alone on penile rehabilitation of erectile dysfunction ED after treatment of post-Robot-Assisted (RA) Radical Prostatectomy (RP) RARP

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≤75 yrs;
* Low-risk PCa (PSA <10 ng/mL and GS <7, ISUP grade 1, and cT1-2a) undergoing nerve sparing RARP;
* preoperative IIEF-5 score ≥ 17;
* First PSA (45d after surgery) <0.2
* compliants patients able to follow the study protocol and fill in IIEF-5 scores and EORTC quality of life questionnaires;
* patients able to provide a written informed consent for the trial.

Exclusion Criteria:

* anaesthesiologic contraindications to robotic surgery;
* patients submitted to pelvic radiotherapy or androgen deprivation;
* patients reporting major postoperative complications (CD≥3);
* cardiovascular contraindications to PDE5i medical treatment.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Impact of LiESWT | 3 years
  To evaluate the impact that the use of low intensity extracorporeal shock waves LiESWT in combination with the early administration of phosphodiesterase 5 inhibitors has on the patient in the process of penile rehabilitation in erectile dysfunction following post-assisted radical prostatectomy robot

SECONDARY OUTCOMES:
Assess how many patients reach orgasm | 3 years
  Compare the rate of patients achieving orgasm. The International Index of Erectile Function short form (IIEF-5) questionnaire is the recognized tool for assessing erectile function both before surgery and during follow-up.
Questionnaires of Quality of life | 3 years
  Compare health-related quality of life outcomes through a validated self-administered questionnaire preoperatively and at postoperative follow-up assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy